CLINICAL TRIAL: NCT05885776
Title: Preoperative Treatment of HR+/HER2+Breast Cancer With Pyrrolitinib Combined With Trastuzumab and AI Efficacy and Safety of: a Single Arm Multicenter Phase II Exploratory Study
Brief Title: Preoperative Treatment of HR+/HER2+Breast Cancer With Pirotinib, Trastuzumab and AI Research
Acronym: PYTHON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tianjin Cancer Hospital
Record Dates: First submitted 2023-03-21; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted combined endocrine therapy (Experimental): Subjects who met the inclusion criteria underwent surgery after 6 cycles of treatment with pyrrolitinib+trastuzumab+AI, and their pathological remission was evaluated after surgery
  Interventions: Drug: Pyrrolidine、trastuzumab、AI

INTERVENTIONS:
Drug: Pyrrolidine、trastuzumab、AI — Subjects who met the inclusion criteria underwent surgery after 6 cycles of treatment with pirotinib+trastuzumab+AI, and their postoperative pathological remission was evaluated.
  Other Names: OFS (OFS includes bilateral eggs Nest removal or GnRHa drugs)

SUMMARY:
Research topic Preoperative efficacy and safety of pyrrolitinib combined with trastuzumab and AI in the treatment of HR+/HER2+breast cancer Overall: A single arm multicenter phase II exploratory study。Subjects HR+/HER2+breast cancer patients in stage Ⅱ~Ⅲ A。

DETAILED DESCRIPTION:
Research topic Preoperative efficacy and safety of pyrrolitinib combined with trastuzumab and AI in the treatment of HR+/HER2+breast cancer Overall: A single arm multicenter phase II exploratory study。Subjects HR+/HER2+breast cancer patients in stage Ⅱ~Ⅲ A。Main research purposes: To explore the efficacy and safety of the combination of large and small molecules (pyrrolidine combined with trastuzumab combined with AI) in the preoperative treatment of early HR+/HER2+breast cancer.Secondary study objective: To explore the feasibility of neoadjuvant descending ladder therapy and the changes in ctDNA to provide clues for screening predictive markers.Primary endpoint: Pathological complete response rate (tpCR: ypT0-is/ypN0)。Secondary end points: optimal overall response rate (BORR), bpCR (ypT0-is), tumor residual load (RCB), disease free survival (DFS), breast retention rate, safety。Pyrrolidine (400mg po qd)，Trastuzumab (initial dose 8 mg/kg, follow-up 6 mg/kg ivgtt, d1, Q 3w, total 6 Period)，Anatriazole (1mg po qd)/ Letrozole (2.5mg po qd).For premenopausal or perimenopausal patients, it is necessary to combine OFS (OFS includes bilateral eggs Nest removal or GnRHa drugs).

ELIGIBILITY:
Inclusion Criteria:

* Female initial treatment patients aged ≥ 18 years and ≤ 75 years old
* ECOG score 0-1
* Stage II-IIIA invasive breast cancer, diameter ≥ 20mm
* HER2 positive (IHC score of 3+, or 2+and ISH test positive)
* ER>10%
* Doctors choose to use letrozole/anastrozole for endocrine therapy
* The definition of menopause includes any of the following: (Previous bilateral oophorectomy; Age)≥ 60 years old; Age<60 years old and without chemotherapy, tamoxifen, toremifen, or ovarian suppressionUnder normal conditions, menopause lasts for ≥ 12 months, and follicle stimulating hormone (FSH) and estradiol are within the postmenopausal range;If receiving tamoxifen or toremifen and age<60 years, FSH and plasma estradiolWithin the postmenopausal range)
* Left ventricular ejection fraction (LVEF) ≥ 50%
* 12 lead electrocardiogram: QT interval (QTcF) corrected by Fridericia method for females<470ms；
* The functional level of the main organs must meet the following requirements: blood routine: ANC ≥ 1.5 × 109/L； PLT≥90 × 109/L； Hb≥90 g/L；Blood biochemistry: TBIL ≤ 2.5 × ULN； ALT and AST ≤ 2.5 × ULN； BUN and Cr ≤ 1.5 × ULN；
* For female subjects who have not undergone menopause or surgical sterilization, during the treatment period and during the study treatment
* Agree to abstain or use effective contraceptive methods for at least 2 months after the next administration; .Volunteer to join this study, sign informed consent, have good compliance, and be willing to cooperate with follow-up.

Exclusion Criteria:

* Stage IIIB-IV or inflammatory breast cancer
* Metastatic tumor
* Previous or concurrent malignant tumors, whose natural history or treatment may interfere with the safety of the research protocol Patients evaluated for sex or efficacy are not eligible to participate in this trial, but basal or squamous cell skin Except for cancer, cervical cancer in situ or bladder cancer, or the subject has no disease (other cancer) to survive At least 5 years.
* Active infections that require systemic treatment
* Has used any medication in this study within 14 days prior to enrollment
* Major surgery (excluding biopsy) performed within 14 days before enrollment
* Gastrointestinal dysfunction or diseases may seriously affect the absorption of drugs in this study (such as ulcerative Disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) or Severe damage to the ability to swallow capsules/tablets
* Known history of myelodysplastic syndrome or acute myeloid leukemia
* Have a history of abdominal fistula, gastrointestinal perforation, or abdominal abscess within 28 days
* Have any history of cerebrovascular accident (CVA) or transient ischemic attack within 12 months
* Within 6 years, there is a history of acute coronary syndrome (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stent implantation) or symptomatic pericarditis

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 48 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Follow up on postoperative pathological reports for evaluation for Pathological complete response rate (tpCR: ypT0-is/ypN0) | 18weeks
  Follow up on postoperative pathological reports for evaluation rely onMiller&Payne principles

SECONDARY OUTCOMES:
Follow up on postoperative pathological reports for evaluation for Optimal overall response rate (BORR) | 18weeks
  Follow up on postoperative pathological reports for evaluation rely onMiller&Payne principles

OTHER OUTCOMES:
Follow up on postoperative pathological reports for evaluation for tumor residual load(RCB) | 18weeks
  Follow up on postoperative pathological reports for evaluation rely on residual cancer burden
Follow up on postoperative pathological reports for evaluation for breast retention rate | 18weeks
  Follow up on postoperative pathological reports for evaluation rely on Number of all breast conserving patients

CONTACTS AND LOCATIONS:
Overall Officials: JIE GE, doctor, Principal Investigator — Tianjin Cancer Hospital
Locations (1):
- Tianjin Cancer Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Patient baseline information, patient safety information
Supporting Information: Study Protocol
Time Frame: March 30, 2025
Access Criteria: Medical scholars in the world